CLINICAL TRIAL: NCT06637670
Title: Acute Effect of Kinesiological Taping on Pain, Quality of Life and Musculoskeletal System Parameters in Individuals with Meniscus Injury: a Randomized, Placebo-Controlled Study
Brief Title: Kinesiological Taping in Individuals with Meniscus Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Kübra Okuyucu, Assistant Professor, Amasya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81180
Record Dates: First submitted 2024-10-03; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2022-07

CONDITIONS: Meniscus Tears
Keywords: kinesiology taping; pain; quality of life; meniscus injury
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomised, placebo-controlled, double-blinded study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The experimental group (Experimental): This group was applied 'Y shaped' kinesiology taping on quadriceps femoris muscle, based on facilitation technique with 25-50% stretching.
  Interventions: Other: Kinesiology taping
- The placebo group (Placebo Comparator): This group was applied a tape without tension, perpendicular to the quadriceps femoris muscle
  Interventions: Other: Placebo taping

INTERVENTIONS:
Other: Kinesiology taping — 'Y shaped' kinesiology taping was applied on quadriceps femoris muscle, based on facilitation technique with 25-50% stretching.
  Arms: The experimental group
Other: Placebo taping — A tape without tension was applied perpendicular on the quadriceps femoris muscle.
  Arms: The placebo group

SUMMARY:
This study aims to explore how kinesiology taping affects people with mild to moderate meniscus injuries (grades I/II), focusing on pain, movement fears, muscle strength, balance, joint movement, and quality of life.

Two groups will be involved: one will receive kinesiology taping on the thigh muscle with some tension, while the other will receive a placebo tape with no tension. Researchers will measure various factors, including pain and muscle strength, both before and 48-72 hours after taping.

DETAILED DESCRIPTION:
This study aims to understand the short-term (acute) effects of kinesiology taping on people with mild to moderate meniscus injuries (grade I/II). These injuries, affecting the cartilage in the knee, can cause pain, reduced mobility, and fear of movement. Kinesiology taping, a popular therapy, involves applying elastic tape to support muscles and joints. This research looked at whether taping could improve pain, muscle strength, movement, balance, and quality of life in patients with these knee injuries.

Study Design The study will use a randomized, placebo-controlled, and double-blinded design, meaning that patients were randomly assigned to two groups, and neither the patients nor the researchers knew which group each person was in during the treatment.

Experimental Group: will receive kinesiology taping on the quadriceps muscle (the large muscle at the front of the thigh) using a 'Y-shaped' technique with moderate tension (25-50% stretch).

Control Group: will receive a placebo tape applied without tension and placed in a different direction.

Measurements

To evaluate the effects of taping, several aspects will be measured both before the tape was applied and 48-72 hours later:

Pain levels Fear of movement (kinesiophobia) Muscle strength (ability to extend the knee) Proprioception (awareness of limb position and force applied) Joint range of motion (how much the knee can bend and straighten) Joint position sense (accuracy in detecting knee position with eyes closed) Quality of life, using a questionnaire (SF-36) that assesses various aspects like physical function and energy levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with meniscus grade I/II,
* Who agreed to participate in the study
* Signed the voluntary consent form

Exclusion Criteria:

* Pregnant individuals
* Individuals with additional knee injuries (e.g., ligament tears) or chronic conditions affecting the knee (e.g., arthritis).
* Patients with grade III meniscus tears or more severe injuries.
* Who had knee surgery in the last 6 months.
* Patients with skin conditions or allergies to adhesive materials or kinesiology tape.
* Individuals with neurological conditions such as multiple sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Pain | Baseline and 48 hours after the application
  Pain assessment was made with Visual Analogue Scale (VAS). The patient was asked to mark where his or her pain was on the scale by writing "0: No pain, 10: Unbearable pain" at the two ends of the 10-centimeter scale.
Knee extension muscle strength | Baseline and 48 hours after the application
  A hand dynamometer (MicroFet 2 HHD) was used to measure the patients' knee extension muscle strength. Measurements were recorded in kilograms. For measurement, the patient was positioned without support, with his legs hanging off the bed from the knees, knees flexed at 90°, feet free and arms crossed over the shoulders. During the measurement, the thigh to be measured was stabilized with one hand after the patients completed maximum knee extension.

SECONDARY OUTCOMES:
Fear of movement | Baseline and 48 hours after the application
  It was evaluated with the Tampa Kinesiophobia Scale (TKÖ). This scale, developed to measure fear of movement/re-injury, consists of 17 questions. The scale includes injury/re-injury and fear-avoidance parameters in work-related activities.
Proprioceptive force sense | Baseline and 48 hours after the application
  It was evaluated with a pressurized biofeedback device. While the patients were lying on the treatment bed in a supine position, the biofeedback device was placed under the knee and its pressure was adjusted to 20 mmHg. Patients were asked to make maximum isometric contraction of the quadriceps femoris muscle and maintain it for 5 seconds. The highest value read from the device during the patients' contractions was recorded.
Joint range of motion | Baseline and 48 hours after the application
  Knee flexion range of motion measurements were made using a goniometer while the patient was lying in the prone position.
Joint position sense | Baseline and 48 hours after the application
  Baseline Digital Inclinometer was used for this. Knee extension movement was performed for the right and left extremities in eyes open and eyes closed positions. The reposition angle method was used to measure joint position sense. According to this method; The patient's extremity was moved to the required position by the physiotherapist. The patient was asked to remember this position by waiting 5 seconds in this position. The patient was then asked to bring his extremity back to that position.
Quality of life | Baseline and 48 hours after the application
  It was evaluated using the SF-36 scale. The scale consists of a total of 36 questions in eight subsections. These sections are: physical function, body pain, limitation due to physical problems, limitation due to emotional problems, cognitive well-being, social competence, energy, general health. In the scale, each section is evaluated separately, and each question is scored between 0 and 100. The increase in score is interpreted as an improvement in health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams S, Whatman C, Hume PA, Sheerin K. Kinesio taping in treatment and prevention of sports injuries: a meta-analysis of the evidence for its effectiveness. Sports Med. 2012 Feb 1;42(2):153-64. doi: 10.2165/11594960-000000000-00000. PMID 22124445
- [Background] Weiss CB, Lundberg M, Hamberg P, DeHaven KE, Gillquist J. Non-operative treatment of meniscal tears. J Bone Joint Surg Am. 1989 Jul;71(6):811-22. PMID 2745476
- [Background] Reicher MA, Hartzman S, Duckwiler GR, Bassett LW, Anderson LJ, Gold RH. Meniscal injuries: detection using MR imaging. Radiology. 1986 Jun;159(3):753-7. doi: 10.1148/radiology.159.3.3754645.
- [Background] Ageberg E. Consequences of a ligament injury on neuromuscular function and relevance to rehabilitation - using the anterior cruciate ligament-injured knee as model. J Electromyogr Kinesiol. 2002 Jun;12(3):205-12. doi: 10.1016/s1050-6411(02)00022-6. PMID 12086815
- [Background] Spindler KP, Schils JP, Bergfeld JA, Andrish JT, Weiker GG, Anderson TE, Piraino DW, Richmond BJ, Medendorp SV. Prospective study of osseous, articular, and meniscal lesions in recent anterior cruciate ligament tears by magnetic resonance imaging and arthroscopy. Am J Sports Med. 1993 Jul-Aug;21(4):551-7. doi: 10.1177/036354659302100412. PMID 8368416